CLINICAL TRIAL: NCT05763381
Title: Photobiomodulation Therapy for Plantar Fasciitis: A Single-Blind Randomized Control Trial
Brief Title: Low-Level Laser Therapy for Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Geneva Foundation (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Musculoskeletal Injury Rehabilitation Research for Operational Readiness (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 222072
Record Dates: First submitted 2023-02-03; First posted 2023-03-10 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-04

CONDITIONS: Plantar Fascitis
Keywords: Plantar Fasciitis; Photobiomodulation Therapy; Tendinopathy; Low Level Laser Therapy
MeSH Terms: conditions — Fasciitis, Plantar; Tendinopathy | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two treatment groups: usual care with PBM therapy, or usual care with sham PBM therapy.
Who Masked: Participant
Masking Description: Single blind masking. The study team knew which group participants were randomized to. Participants did not know which group they were in until after 6 week follow up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- The Usual Care + PBM Group (Active Comparator): Participants that are assigned to this group will receive active treatment with PBM 3 times a week for 3 weeks for a total of 9 treatments.
  Interventions: Device: Photobiomodulation Therapy (PBMT)
- The Usual Care + Sham (Placebo) PBM Group (Placebo Comparator): Participants that are assigned to this group will receive Sham PBM therapy 3 times a week for 3 weeks for a total of 9 treatments. Sham PBM therapy is an inactive harmless treatment that is intended to mimic the active PBM treatment.
  At the completion of the initial 6 weeks, the Usual Care + Sham (Placebo) PBM Group will be unblinded, and may choose to cross-over and complete another 6 weeks in the active treatment group. If participants choose to cross-over and receive active PBMT, they will re-complete all of the original study procedures (with the exception of screening, as participants have qualified for the study, and baseline data collection, as the study team will use the 6-week follow-up data as the new baseline prior to active PBMT treatment.
  Interventions: Device: Sham-Photobiomodualtion Therapy (Sham-PBMT)

INTERVENTIONS:
Device: Photobiomodulation Therapy (PBMT) — Participants will receive PBMT with the PBM device over the course of three consecutive weeks (three treatments per week). PBM treatments will take approximately 5-10 minutes to administer at each session. Specific treatment parameters will be based on measurements of calf, ankle, and foot using pre-calculated treatment tables; participants will receive 10 J/cm2, 25W output power, and the length of the treatment will be dependent on treatment area (size). PBMT will be administered by a trained member of the study team using the LightForce® XPi therapy laser, provided by LiteCure, LLC/DJO Global (New Castle, DE). The LightForce® XPi therapy laser is an FDA cleared device for the treatment of pain. The trained team members will use the Smart Hand Piece technology, which achieves effective treatments and improves dosing accuracy by assessing the operator's speed and providing real-time visual (red - amber - green light) and sensory feedback.
  Arms: The Usual Care + PBM Group
Device: Sham-Photobiomodualtion Therapy (Sham-PBMT) — Sham-PBM treatment time will be calculated in the same way as the PBM treatment group, with the time of treatment dependent on the size of the treatment area. The sham-PBMT will be administered by rolling the massage ball over the plantar surface of the foot and dorsal aspect of the calf in contact with the participants' skin. Because emission of photons at the selected treatment parameters may cause participants in the treatment group to feel warmth, the massage ball will be warmed in the sham-PBMT. The device will be turned on, so the red aiming beam will be visible, but the operator will not activate the switch to emit photons.
  Arms: The Usual Care + Sham (Placebo) PBM Group

SUMMARY:
Plantar fasciitis (PF), a degenerative injury of the connective tissue in the foot, results in pain-related disability in Service Members and contributes to decreased physical activity and excessive healthcare costs. Even if effective, current treatment protocols may require 6-12 months of therapy to return individuals to pain-free activity. Photobiomodulation therapy (PBMT) uses non-ionizing light to elicit biological changes in tissues resulting in beneficial therapeutic outcomes. Evidence supports use of PBM for other degenerative connective tissue conditions, such as achilles tendinopathy and epicondylitis. A previous pilot study was completed in an active-duty military and civilian population, which demonstrated a positive effect of two PBM dose parameters on function and pain levels in participants with chronic PF when combined with stretching and ice. These positive findings from the aforementioned study are promising in the treatment of this common and debilitating issue, but require the addition of a sham comparison to rigorously eliminate any potential placebo effect of the treatment protocol, and further refine the treatment protocol in order to make evidence-based clinical recommendations. As such, proposing a follow-up study and the addition of an objective outcome measure will strengthen the impact of the study.

SPECIFIC AIM 1: To assess the clinical effectiveness of photobiomodulation compared to sham photobiomodulation to improve function and decrease pain.

SPECIFIC AIM 2: To evaluate the effectiveness of photobiomodulation compared to sham photobiomodulation to resolve plantar fascial thickening. DESIGN: A prospective randomized sham-controlled trial to meet the aims of the study.

METHOD: A sample of up to 100 active-duty military members will be randomly assigned to the Sham-PBMT or PBMT group. At baseline, during the treatment protocol, and at long-term (3 and 6 months) follow-up, measures of foot function, pain, and plantar fascial thickness will be collected for analysis. The proposed methods will allow the study team to establish if PBMT is clinically effective to accelerate recovery compared to Sham-PBMT and result in resolution of fascial thickening, decrease in pain, and improved function.

LONG-TERM GOAL: The long-term goals of the research include developing PBMT protocols for broad application to other painful and duty-limiting conditions.

DETAILED DESCRIPTION:
Recruitment, Pre-Screening (before consent), Study Introduction & Informed Consent:

Potential participants will be identified via four methods:

1. Under the provisions of the Partial HIPAA Waiver, local study providers will review medical records of patients coming into the Orthopedic and Podiatry Clinics for suspected plantar fasciitis to identify prospective research participants for the purposes of seeking their authorization to participate/use their protected health information for this research study. In these cases, the study team will receive approval from the potential participant's provider prior to approaching for possible study participation.
2. Direct referral from local healthcare providers in the local Family Medicine, Podiatry, Physical Therapy, and Physical Medicine & Rehabilitation (PM&R) clinics.
3. Patients may self-refer to participate in the study. Interested potential participants will be able to contact a member of the study team via phone or email. Potential participants who contact the study team directly will be instructed to access the Physical Therapy clinic or their primary care manager for a physical exam and diagnosis of Plantar Fasciitis (PF) or confirmation of a previous PF diagnosis.
4. Study advertisements will be posted, and copies will be provided to clinic staff.

Eligibility will be determined in person. If the potential participant meets eligibility criteria as determined by the Inclusion/Exclusion CRF and expresses interest in participating, an authorized study team member will initiate the formal consent discussion and, if applicable, obtain informed consent.

Baseline Data Collection (post-consent): Prior to receiving the assigned study treatment, participants will provide their contact information and complete a series of baseline outcome measures (Demographics CRF and Baseline Data Collection CRF) and have their plantar fascia thickness measured within the Podiatry clinic. A study team member will also acquire measurements of the participant's calf, ankle, and foot to calculate the appropriate PBMT dose.

Randomization: Participants will be randomly assigned to a study group (PBMT+UC or Sham PBMT+UC) using a computer-generated randomization model prepared by the study biostatistician.

Study Treatments (PBMT+UC or Sham PBMT+UC): All participants, regardless of study arm assignment, will be asked to complete the UC Protocol, which consists of a daily regimen of stretching and cryotherapy that includes 3-5 minutes of stretching upon waking, then approximately 3-5 minutes of stretching and 3-5 minutes of cryotherapy throughout the day, for the duration of 6 weeks.

Participants will receive PBMT or sham-PBMT with the PBM device over the course of three consecutive weeks (three treatments per week). PBM treatments will take approximately 5-10 minutes to administer at each session. Specific treatment parameters will be based on measurements of calf, ankle, and foot using pre-calculated treatment tables; participants will receive 10 J/cm2, 25W output power, and the length of the treatment will be dependent on the treatment area (size).

Photobiomodulation Therapy (PBMT): PBMT will be administered by a trained member of the study team using the LightForce® XPi therapy laser, provided by LiteCure, LLC/DJO Global (New Castle, DE). The LightForce® XPi therapy laser is an FDA cleared device for the treatment of pain. The trained team members will use the Smart Hand Piece technology, which achieves effective treatments and improves dosing accuracy by assessing the operator's speed and providing real-time visual (red - amber - green light) and sensory feedback. The Smart Hand Piece is calibrated to shutoff when moving too slowly, and warn the operator when moving too fast by vibrating. The therapy is delivered through a flexible optical fiber threaded through the hand piece, which contains a rolling sapphire massage ball. The PBM therapy will be administered by rolling the massage ball over the plantar surface of the foot and dorsal aspect of the calf in contact with the participants' skin.

Sham-Photobiomodulation Therapy (Sham-PBMT): Sham-PBM treatment time will be calculated in the same way as the PBM treatment group, with the time of treatment dependent on the size of the treatment area. The sham-PBMT will be administered by rolling the massage ball over the plantar surface of the foot and dorsal aspect of the calf in contact with the participants' skin. Because emission of photons at the selected treatment parameters may cause participants in the treatment group to feel warmth, the massage ball will be warmed in the sham-PBMT. The device will be turned on, so the red aiming beam will be visible, but the operator will not activate the switch to emit photons. The following safeguards will be in place to prevent exposure to PBM and potential unexpected crossover or protocol deviations, as follows:

The PBM device requires multiple steps to emit photons. The device first must be powered on, then settings are selected (in this case, power will be 25 watts, and the time will be determined by the algorithm based on the treatment area measurements). Next, there is a 'standby' button that is activated on the touch screen, and finally, there is a finger switch on the handpiece that must be pressed to initiate the treatment. There is a beep that sounds for the duration of the active treatment.

For the sham condition, the device will be turned on and the settings will be selected, but the standby button and the finger switch on the handpiece will not be activated. This way, there is no chance that the device will be emitting photons. Since the device will not emit active treatment, there will not be a beeping sound from the device; this beeping noise will be replicated in another way for the sham-PBMT. At the completion of the initial 6 weeks, Sham-PBMT participants will be unblinded, and may choose to cross-over and complete another 6 weeks in the active treatment group. If Sham-PBMT participants choose to cross-over and receive active PBMT, participants will re-complete all of the original study procedures (with the exception of screening).

Follow Up Data Collection: In addition to their 3x weekly for 3 weeks PBM or Sham-PBM treatments, participants will report to the study team in person approximately 3 weeks (+/- 3 days) and 6 weeks (+/- 3 days) after the start of their PBM or Sham-PBM treatment to complete the follow-up questionnaires, turn in their Pain Diary, and undergo ultrasound imaging to measure changes in plantar fascia thickness at 3-weeks and 6-weeks.

Long-term follow up questionnaires will be captured remotely (e.g., entered directly into REDCap using a personalized coded link with no log-in required, verbally over the phone with a study team member, etc.) at approximately 3-months (+/- 10 days/weeks) post-start of PBM treatment. For Sham-PBMT participants who cross-over, their 3-month follow-up will be timed from the first day of their active PBM treatment, not their Sham-PBM treatment. Reminder phone calls and emails will be sent to participants at the phone and email address provided to the study team before the 3-month follow-up time point. Participants will be evaluated for adverse events at each follow-up time point and any complications will be documented.

Study participation ends after the 3-month follow-up research activities are completed. Participants initially randomized to the PBMT group will participate in the study for approximately 3 months. Participants initially assigned to the Sham-PBMT group who choose to cross-over and receive active PBMT post-unblinding will be in the study for approximately 4.5 months total.

Ultrasound Measurement: Plantar fascia thickness will be measured by an MSK US trained provider utilizing an ultrasound system. The participant will be identified on the ultrasound system using only the assigned participant ID. The patient will be positioned prone on an examination table with the leg extending off the end so the foot projects downward in a relaxed state. Using a linear transducer for best resolution, the plantar fascia will be evaluated in the long axis to determine the site to be measured as identified by the bony contour demonstrated. The vertical thickness of the plantar fascia will be documented in both long and short axis at this point. The points measured will be from the edge of the bone to the outer layer of the plantar fascia.

Plantar fascia thickness will be measured in two orthogonal planes (90 degrees different - long axis and short axis of the structure) at the site identified by the bone contour. The measurement will be conducted by MSK US trained providers, either in Physical Therapy or Physical Medicine and Rehab clinics.

ELIGIBILITY:
Inclusion Criteria:

* DEERS eligible
* Able to read and understand English language for consent purposes
* Experience pain in the bottom of foot and/or heel at any time during the day
* Diagnosis of Plantar Fasciitis (PF) by a healthcare provider based on accepted diagnostic criteria
* Abel to commit to study procedures, including a 6-week intervention and 3 month follow-up
* Have experienced symptoms of PF for at least 3 months

Exclusion Criteria:

* Diagnosed with a calcaneal (heel) fracture by a healthcare provider
* Currently pregnant or plan to become pregnant during intervention period (safety of PBM not established in pregnancy)
* History of traumatic injury to symptomatic foot/feet
* Previous surgery, or other invasive treatment for same condition
* Significant portion of calf area covered in tattoos/ink/scarring (pigment in ink can absorb light, causing overheating of skin)
* History of neuropathy or inability to detect changes in skin temperature (increased risk of skin warming due to inability to detect change)
* Current use of medications associated with sensitivity to heat or light (e.g., amiodarone, chlorpromazine, doxycycline, hydrochlorothiazide, nalidixic acid, naproxen, piroxicam, tetracycline, thioridazine, voriconazole)
* Concurrent participation in another research study addressing pain issue
* Current use of pacemaker
* Current or chronic sciatica resulting in chronic or intermittent lower extremity pain, numbness, or tingling
* Previous enrollment in this study for contralateral foot

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Any research data shared with an approved agency for review will be linked only to the participant's unique study ID and not with the personal identity of the participant. If the research data is used in scholarly presentations or journal articles, the investigators will protect the anonymity of individual participants and report only aggregate data where appropriate. Participants will not be individually identified in any publication or presentation of research results.
Supporting Information: ICF
Time Frame: De-identified research data will be shared with Military Injury Rehabilitation Research for Operational Readiness (MIRROR) and maintained indefinitely for possible use in future research.
Access Criteria: De-identified data will only be accessible by authorized study team members and oversight officials, the local Madigan Human Research Protections Office, the IRB, authorized staff from USU, and authorized staff from Musculoskeletal Injury Rehabilitation Research for Operational Readiness, which is based out of the department of Physical Medicine & Rehabilitation at USU, and is serving as the data coordinator.

REFERENCES:
- [Background] Scher DL, Belmont PJ Jr, Bear R, Mountcastle SB, Orr JD, Owens BD. The incidence of plantar fasciitis in the United States military. J Bone Joint Surg Am. 2009 Dec;91(12):2867-72. doi: 10.2106/JBJS.I.00257. PMID 19952249
- [Background] Dyck DD Jr, Boyajian-O'Neill LA. Plantar fasciitis. Clin J Sport Med. 2004 Sep;14(5):305-9. doi: 10.1097/00042752-200409000-00010. No abstract available. PMID 15377971
- [Background] Rosenbaum AJ, DiPreta JA, Misener D. Plantar heel pain. Med Clin North Am. 2014 Mar;98(2):339-52. doi: 10.1016/j.mcna.2013.10.009. Epub 2013 Dec 10. PMID 24559879
- [Background] DiGiovanni BF, Nawoczenski DA, Lintal ME, Moore EA, Murray JC, Wilding GE, Baumhauer JF. Tissue-specific plantar fascia-stretching exercise enhances outcomes in patients with chronic heel pain. A prospective, randomized study. J Bone Joint Surg Am. 2003 Jul;85(7):1270-7. doi: 10.2106/00004623-200307000-00013. PMID 12851352
- [Background] Schwartz EN, Su J. Plantar fasciitis: a concise review. Perm J. 2014 Winter;18(1):e105-7. doi: 10.7812/TPP/13-113. PMID 24626080
- [Background] Franceschi F, Papalia R, Paciotti M, Franceschetti E, Di Martino A, Maffulli N, Denaro V. Obesity as a risk factor for tendinopathy: a systematic review. Int J Endocrinol. 2014;2014:670262. doi: 10.1155/2014/670262. Epub 2014 Aug 19. PMID 25214839
- [Background] Roy TC. Diagnoses and mechanisms of musculoskeletal injuries in an infantry brigade combat team deployed to Afghanistan evaluated by the brigade physical therapist. Mil Med. 2011 Aug;176(8):903-8. doi: 10.7205/milmed-d-11-00006. PMID 21882780
- [Background] Roy TC, Knapik JJ, Ritland BM, Murphy N, Sharp MA. Risk factors for musculoskeletal injuries for soldiers deployed to Afghanistan. Aviat Space Environ Med. 2012 Nov;83(11):1060-6. doi: 10.3357/asem.3341.2012. PMID 23156094
- [Background] Cameron KL, Owens BD. The burden and management of sports-related musculoskeletal injuries and conditions within the US military. Clin Sports Med. 2014 Oct;33(4):573-89. doi: 10.1016/j.csm.2014.06.004. PMID 25280610
- [Background] Lemont H, Ammirati KM, Usen N. Plantar fasciitis: a degenerative process (fasciosis) without inflammation. J Am Podiatr Med Assoc. 2003 May-Jun;93(3):234-7. doi: 10.7547/87507315-93-3-234. PMID 12756315
- [Background] Orchard J. Plantar fasciitis. BMJ. 2012 Oct 10;345:e6603. doi: 10.1136/bmj.e6603. No abstract available. PMID 23054045
- [Background] Franceschi F, Papalia R, Franceschetti E, Paciotti M, Maffulli N, Denaro V. Platelet-rich plasma injections for chronic plantar fasciopathy: a systematic review. Br Med Bull. 2014 Dec;112(1):83-95. doi: 10.1093/bmb/ldu025. Epub 2014 Sep 19. PMID 25239050
- [Background] Hammer WI. The effect of mechanical load on degenerated soft tissue. J Bodyw Mov Ther. 2008 Jul;12(3):246-56. doi: 10.1016/j.jbmt.2008.03.007. Epub 2008 Jun 3. PMID 19083680
- [Background] Tountas AA, Fornasier VL. Operative treatment of subcalcaneal pain. Clin Orthop Relat Res. 1996 Nov;(332):170-8. doi: 10.1097/00003086-199611000-00023. PMID 8913160
- [Background] Miller LE, Latt DL. Chronic Plantar Fasciitis is Mediated by Local Hemodynamics: Implications for Emerging Therapies. N Am J Med Sci. 2015 Jan;7(1):1-5. doi: 10.4103/1947-2714.150080. PMID 25709971
- [Background] Jones BH, Canham-Chervak M, Canada S, Mitchener TA, Moore S. Medical surveillance of injuries in the u.s. Military descriptive epidemiology and recommendations for improvement. Am J Prev Med. 2010 Jan;38(1 Suppl):S42-60. doi: 10.1016/j.amepre.2009.10.014. PMID 20117600
- [Background] Canyilmaz E, Canyilmaz F, Aynaci O, Colak F, Serdar L, Uslu GH, Aynaci O, Yoney A. Prospective Randomized Comparison of the Effectiveness of Radiation Therapy and Local Steroid Injection for the Treatment of Plantar Fasciitis. Int J Radiat Oncol Biol Phys. 2015 Jul 1;92(3):659-66. doi: 10.1016/j.ijrobp.2015.02.009. Epub 2015 Apr 28. PMID 25936814
- [Background] Rompe JD. Plantar fasciopathy. Sports Med Arthrosc Rev. 2009 Jun;17(2):100-4. doi: 10.1097/JSA.0b013e3181a3d60e. PMID 19440137
- [Background] Anders JJ, Lanzafame RJ, Arany PR. Low-level light/laser therapy versus photobiomodulation therapy. Photomed Laser Surg. 2015 Apr;33(4):183-4. doi: 10.1089/pho.2015.9848. No abstract available. PMID 25844681
- [Background] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511
- [Background] Alghadir A, Omar MT, Al-Askar AB, Al-Muteri NK. Effect of low-level laser therapy in patients with chronic knee osteoarthritis: a single-blinded randomized clinical study. Lasers Med Sci. 2014 Mar;29(2):749-55. doi: 10.1007/s10103-013-1393-3. Epub 2013 Aug 3. PMID 23912778
- [Background] Chow RT, Johnson MI, Lopes-Martins RA, Bjordal JM. Efficacy of low-level laser therapy in the management of neck pain: a systematic review and meta-analysis of randomised placebo or active-treatment controlled trials. Lancet. 2009 Dec 5;374(9705):1897-908. doi: 10.1016/S0140-6736(09)61522-1. Epub 2009 Nov 13. PMID 19913903
- [Background] Tumilty S, McDonough S, Hurley DA, Baxter GD. Clinical effectiveness of low-level laser therapy as an adjunct to eccentric exercise for the treatment of Achilles' tendinopathy: a randomized controlled trial. Arch Phys Med Rehabil. 2012 May;93(5):733-9. doi: 10.1016/j.apmr.2011.08.049. PMID 22541305
- [Background] Tumilty S, Munn J, Abbott JH, McDonough S, Hurley DA, Baxter GD. Laser therapy in the treatment of achilles tendinopathy: a pilot study. Photomed Laser Surg. 2008 Feb;26(1):25-30. doi: 10.1089/pho.2007.2126. PMID 18248158
- [Background] Tumilty S, Munn J, McDonough S, Hurley DA, Basford JR, Baxter GD. Low level laser treatment of tendinopathy: a systematic review with meta-analysis. Photomed Laser Surg. 2010 Feb;28(1):3-16. doi: 10.1089/pho.2008.2470. PMID 19708800
- [Background] Haslerud S, Magnussen LH, Joensen J, Lopes-Martins RA, Bjordal JM. The efficacy of low-level laser therapy for shoulder tendinopathy: a systematic review and meta-analysis of randomized controlled trials. Physiother Res Int. 2015 Jun;20(2):108-25. doi: 10.1002/pri.1606. Epub 2014 Dec 2. PMID 25450903
- [Background] Oliveira FS, Pinfildi CE, Parizoto NA, Liebano RE, Bossini PS, Garcia EB, Ferreira LM. Effect of low level laser therapy (830 nm) with different therapy regimes on the process of tissue repair in partial lesion calcaneous tendon. Lasers Surg Med. 2009 Apr;41(4):271-6. doi: 10.1002/lsm.20760. PMID 19347936
- [Background] Ng GY, Fung DT. The combined treatment effects of therapeutic laser and exercise on tendon repair. Photomed Laser Surg. 2008 Apr;26(2):137-41. doi: 10.1089/pho.2007.2145. PMID 18341419
- [Background] Basford JR, Malanga GA, Krause DA, Harmsen WS. A randomized controlled evaluation of low-intensity laser therapy: plantar fasciitis. Arch Phys Med Rehabil. 1998 Mar;79(3):249-54. doi: 10.1016/s0003-9993(98)90002-8. PMID 9523774
- [Background] Jastifer JR, Catena F, Doty JF, Stevens F, Coughlin MJ. Low-Level Laser Therapy for the Treatment of Chronic Plantar Fasciitis: A Prospective Study. Foot Ankle Int. 2014 Jun;35(6):566-571. doi: 10.1177/1071100714523275. PMID 24510123
- [Background] Macias DM, Coughlin MJ, Zang K, Stevens FR, Jastifer JR, Doty JF. Low-Level Laser Therapy at 635 nm for Treatment of Chronic Plantar Fasciitis: A Placebo-Controlled, Randomized Study. J Foot Ankle Surg. 2015 Sep-Oct;54(5):768-72. doi: 10.1053/j.jfas.2014.12.014. Epub 2015 Mar 10. PMID 25769363
- [Background] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Background] Buckenmaier CC 3rd, Galloway KT, Polomano RC, McDuffie M, Kwon N, Gallagher RM. Preliminary validation of the Defense and Veterans Pain Rating Scale (DVPRS) in a military population. Pain Med. 2013 Jan;14(1):110-23. doi: 10.1111/j.1526-4637.2012.01516.x. Epub 2012 Nov 8. PMID 23137169
- [Background] Nassif TH, Hull A, Holliday SB, Sullivan P, Sandbrink F. Concurrent Validity of the Defense and Veterans Pain Rating Scale in VA Outpatients. Pain Med. 2015 Nov;16(11):2152-61. doi: 10.1111/pme.12866. Epub 2015 Aug 8. PMID 26257151
- [Background] Tumilty S, Mani R, Baxter GD. Photobiomodulation and eccentric exercise for Achilles tendinopathy: a randomized controlled trial. Lasers Med Sci. 2016 Jan;31(1):127-35. doi: 10.1007/s10103-015-1840-4. Epub 2015 Nov 26. PMID 26610637
- [Background] Redberg RF. Sham controls in medical device trials. N Engl J Med. 2014 Sep 4;371(10):892-3. doi: 10.1056/NEJMp1406388. No abstract available. PMID 25184861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 71 consented to participate in the study.
Pre-assignment Details: 71 participants consented, 2 were withdrawn prior to randomization (1 self-withdrawal, 1 withdrawn by PI). 69 were randomized to the study treatments.
Groups:
- The Usual Care + PBM Group: Participants that are assigned to this group will receive active treatment with PBM 3 times a week for 3 weeks for a total of 9 treatments.
  Photobiomodulation Therapy (PBMT): Participants will receive PBMT with the PBM device over the course of three consecutive weeks (three treatments per week). PBM treatments will take approximately 5-10 minutes to administer at each session. Specific treatment parameters will be based on measurements of calf, ankle, and foot using pre-calculated treatment tables; participants will receive 10 J/cm2, 25W output power, and the length of the treatment will be dependent on treatment area (size).
  PBMT will be administered by a trained member of the study team using the LightForce® XPi therapy laser, provided by LiteCure, LLC/DJO Global (New Castle, DE). The LightForce® XPi therapy laser is an FDA cleared device for the treatment of pain. The trained team members will use the Smart Hand Piece technology, which achieves effective treatments and improves dosing accuracy by assessing the operator's speed and providing real-time visual (red - amber - green light) and sensory feedback.
- The Usual Care + Sham (Placebo) PBM Group: Participants that are assigned to this group will receive Sham PBM therapy 3 times a week for 3 weeks for a total of 9 treatments. Sham PBM therapy is an inactive harmless treatment that is intended to mimic the active PBM treatment.
  Sham-Photobiomodualtion Therapy (Sham-PBMT): Sham-PBM treatment time will be calculated in the same way as the PBM treatment group, with the time of treatment dependent on the size of the treatment area. The sham-PBMT will be administered by rolling the massage ball over the plantar surface of the foot and dorsal aspect of the calf in contact with the participants' skin. Because emission of photons at the selected treatment parameters may cause participants in the treatment group to feel warmth, the massage ball will be warmed in the sham-PBMT. The device will be turned on, so the red aiming beam will be visible, but the operator will not activate the switch to emit photons.
  At the completion of the initial 6 weeks, the Usual Care + Sham (Placebo) PBM Group will be unblinded, and may choose to cross-over and complete another 6 weeks in the active treatment group. If participants choose to cross-over and receive active PBMT, they will re-complete all of the original study procedures (with the exception of screening, as participants have qualified for the study, and baseline data collection, as the study team will use the 6-week follow-up data as the new baseline prior to active PBMT treatment.
Period: Overall Study
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Started | 34 | 35
Cross-over to Intervention | 0 | 26
Completed | 31 | 30
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: 2 participants withdrew from the study prior to randomization and 69 randomized participants were analyzed for baseline characteristics.
Groups:
- The Usual Care + PBM Group: Participants that were assigned to this group received active treatment with PBM 3 times a week for 3 weeks for a total of 9 treatments.
  Photobiomodulation Therapy (PBMT): Participants received PBMT with the PBM device over the course of three consecutive weeks (three treatments per week). PBM treatments took approximately 5-10 minutes to administer at each session. Specific treatment parameters were based on measurements of calf, ankle, and foot using pre-calculated treatment tables; participants received receive 10 J/cm2, 25W output power, and the length of the treatment was dependent on treatment area (size).
  PBMT was administered by a trained member of the study team using the LightForce® XPi therapy laser, provided by LiteCure, LLC/DJO Global (New Castle, DE). The LightForce® XPi therapy laser is an FDA cleared device for the treatment of pain. The trained team members used the Smart Hand Piece technology, which achieves effective treatments and improves dosing accuracy by assessing the operator's speed and providing real-time visual (red - amber - green light) and sensory feedback.
- The Usual Care + Sham (Placebo) PBM Group: Participants that were assigned to this group received Sham PBM therapy 3 times a week for 3 weeks for a total of 9 treatments. Sham PBM therapy was an inactive harmless treatment that was intended to mimic the active PBM treatment.
  Sham-Photobiomodualtion Therapy (Sham-PBMT): Sham-PBM treatment time was calculated in the same way as the PBM treatment group, with the time of treatment dependent on the size of the treatment area. The sham-PBMT was administered by rolling the massage ball over the plantar surface of the foot and dorsal aspect of the calf in contact with the participants' skin. Because emission of photons at the selected treatment parameters may cause participants in the treatment group to feel warmth, the massage ball was warmed in the sham-PBMT. The device was turned on to make the red aiming beam visible, but the operator did not activate the switch to emit photons.
- Total: Total of all reporting groups
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 35 | 69
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 24 | 25 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 9 | 7 | 16
  Black or African American | 4 | 4 | 8
  White(Not Hispanic) | 14 | 14 | 28
  Hispanic | 7 | 8 | 15
  Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Foot and Ankle Ability Measure (FAAM)
Description: The FAAM is a 29-item self-report instrument that assesses physical function in foot and ankle impairments which included PF cases in development. There are two subscales, Activities of Daily Living(ADL) (21- item) and Sports (7-item). Each item is scored on a 5-point Likert scale (4='no difficulty at all' to 0='unable to do'); points are transformed to a percentage (100%=no dysfunction). The minimum clinically important difference 8 & 9 points for ADL & Sports subscale, respectively. Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction and 0% being dysfunction.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percentage of function
Groups:
- The Usual Care + PBM Group: Participants that were assigned to this group received treatment with PBM 3 times a week for 3 weeks for a total of 9 treatments.
  Photobiomodulation Therapy (PBMT): Participants received PBMT with the PBM device over the course of three consecutive weeks (three treatments per week). PBM treatments took approximately 5-10 minutes to administer at each session. Specific treatment parameters were based on measurements of calf, ankle, and foot using pre-calculated treatment tables; participants received 10 J/cm2, 25W output power, and the length of the treatment was dependent on treatment area (size).
  PBMT was administered by a trained member of the study team using the LightForce® XPi therapy laser, provided by LiteCure, LLC/DJO Global (New Castle, DE). The LightForce® XPi therapy laser is an FDA cleared device for the treatment of pain. The trained team members used the Smart Hand Piece technology, which achieves effective treatments and improves dosing accuracy by assessing the operator's speed and providing real-time visual (red - amber - green light) and sensory feedback.
- The Usual Care + Sham (Placebo) PBM Group: Participants that were assigned to this group received Sham PBM therapy 3 times a week for 3 weeks for a total of 9 treatments. Sham PBM therapy was an inactive harmless treatment that was intended to mimic the active PBM treatment.
  Sham-Photobiomodualtion Therapy (Sham-PBMT): Sham-PBM treatment time will be calculated in the same way as the PBM treatment group, with the time of treatment dependent on the size of the treatment area. The sham-PBMT was administered by rolling the massage ball over the plantar surface of the foot and dorsal aspect of the calf in contact with the participants' skin. Because emission of photons at the selected treatment parameters may cause participants in the treatment group to feel warmth, the massage ball was warmed in the sham-PBMT. The device was turned on to make the red aiming beam visible, but the operator did not activate the switch to emit photons.
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 34 | 35
Percentage of function
  Activities of Daily Living (21- item) | 47.00 (13.97) | 45.28 (12.42)
  Sports (7-item) | 11.65 (5.84) | 11.72 (6.29)

2. Primary Outcome: Foot and Ankle Ability Measure (FAAM)
Description: as for outcome 1
Time Frame: 3-Week
Population: 64 enrolled participants were analyzed for 3-week follow-up results. 3 participants that were assigned to the Usual Care + PBM Group and 2 participants that were assigned to the Usual Care + Sham (Placebo) PBM Group withdrew from the study prior to 3-week follow-up.
Measure: Mean (Standard Deviation); unit: Percentage of function
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 31 | 33
Percentage of function
  Activities of Daily Living (21- item) | 54.00 (11.82) | 53.79 (12.68)
  Sports (7-item) | 15.42 (5.91) | 13.27 (6.72)

3. Primary Outcome: Foot and Ankle Ability Measure (FAAM)
Description: as for outcome 1
Time Frame: 6-week
Population: 62 enrolled participants completed 6-week follow-up and were analyzed for 6-week follow-up results. 2 participants that were assigned to the Usual Care + Sham (Placebo) PBM Group withdrew from the study prior to 6-week follow-up.
Measure: Mean (Standard Deviation); unit: Percentage of function
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 31 | 31
Percentage of function
  Activities of Daily Living (21- item) | 56.81 (14.79) | 53.26 (14.64)
  Sports (7-item) | 17.84 (6.60) | 13.58 (7.06)

4. Primary Outcome: Foot and Ankle Ability Measure (FAAM)
Description: as for outcome 1
Time Frame: 3-month
Population: 31 participants from the Usual Care + PBM Group and 4 participants from the Usual Care + Sham (Placebo) PBM Group completed 3-month randomized followed up. 26 randomized participants from the Usual Care + Sham (Placebo) PBM Group crossed over at 6-week follow-up and received the study intervention.
Measure: Mean (Standard Deviation); unit: Percentage of function
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 31 | 4
Percentage of function
  Activities of Daily Living (21- item) | 58.29 (18.06) | 52.00 (18.69)
  Sports (7-item) | 17.35 (8.49) | 10.75 (8.17)

5. Primary Outcome: Pain Diary Defense and Veterans Pain Rating Scale (DVPRS)
Description: Defense and Veterans Pain Rating Scale (DVPRS) 72. The 5-item scale integrates a numeric pain rating scale with visual facial cues and word descriptors as well as 4 supplemental questions on pain interference.
  Rating scale from 0-10 (0=No pain, 10=As bad as it could be nothing else matters); higher score equal worse outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pain units on a scale
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 34 | 35
pain units on a scale | 4.97 (2.09) | 5.17 (1.85)

6. Primary Outcome: Pain Diary Defense and Veterans Pain Rating Scale (DVPRS)
Description: as for outcome 5
Time Frame: 3-Week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pain units on a scale
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 31 | 33
pain units on a scale | 4.19 (2.09) | 4.03 (1.83)

7. Primary Outcome: Pain Diary Defense and Veterans Pain Rating Scale (DVPRS)
Description: as for outcome 5
Time Frame: 6-Week
Population: 62 enrolled participants were analyzed for 6-week follow-up results. 2 participants that were assigned to the Usual Care + Sham (Placebo) PBM Group withdrew from the study prior to 6-week follow-up.
Measure: Mean (Standard Deviation); unit: pain units on a scale
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 31 | 31
pain units on a scale | 3.71 (1.99) | 4.00 (2.05)

8. Primary Outcome: Pain Diary Defense and Veterans Pain Rating Scale (DVPRS)
Description: as for outcome 5
Time Frame: 3-Month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pain units on a scale
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 33 | 26
pain units on a scale | 3.47 (2.60) | 4.50 (3.20)

9. Primary Outcome: Ultrasound Measurement (Plantar Fascial Thickness)
Description: Plantar fascia thickness was measured by an MSK US trained provider utilizing an ultrasound system. The patient was positioned prone on an examination table with the leg extending off the end so the foot projects downward in a relaxed state. Using a linear transducer for best resolution, the plantar fascia was evaluated in the long axis to determine the site to be measured as identified by the bony contour. The vertical thickness of the plantar fascia will be documented in both long and short axis at this point. The points measured were from the edge of the bone to the outer layer of the plantar fascia. The average of both long and short-axis measurements was analyzed for the PF thinness results.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 34 | 35
millimeters | 4.18 (1.98) | 4.29 (1.23)

10. Primary Outcome: Ultrasound Measurement (Plantar Fascial Thickness)
Description: as for outcome 9
Time Frame: 3-Week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 31 | 33
millimeters | 3.955 (1.24) | 4.375 (1.165)

11. Primary Outcome: Ultrasound Measurement (Plantar Fascial Thickness)
Description: as for outcome 9
Time Frame: 6-Week
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group
Number analyzed (Participants) | 31 | 31
millimeters | 4.155 (1.825) | 4.665 (1.045)

12. Other Pre Specified Outcome: Foot and Ankle Ability Measure (FAAM)
Description: as for outcome 1
Time Frame: 3-Week Cross-over
Measure: Mean (Standard Deviation); unit: Percentage of function
Groups:
- The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention: Participants that were decided to cross-over to this group received active treatment with PBM 3 times a week for 3 weeks for a total of 9 treatments.
  Photobiomodulation Therapy (PBMT): Participants received PBMT with the PBM device over the course of three consecutive weeks (three treatments per week). PBM treatments took approximately 5-10 minutes to administer at each session. Specific treatment parameters were based on measurements of calf, ankle, and foot using pre-calculated treatment tables; participants received 10 J/cm2, 25W output power, and the length of the treatment dependent on treatment area (size).
  PBMT was administered by a trained member of the study team using the LightForce® XPi therapy laser, provided by LiteCure, LLC/DJO Global (New Castle, DE). The LightForce XPi therapy laser is an FDA cleared device for the treatment of pain. The trained team member used the Smart Hand Piece technology, which achieves effective treatments and improves dosing accuracy by assessing the operator's speed and providing real-time visual (red - amber - green light) and sensory feedback.
Arm/Group | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention
Number analyzed (Participants) | 26
Percentage of function
  Activities of Daily Living (21- item) | 57.07 (14.88)
  Sports (7-item) | 16.11 (7.92)

13. Other Pre Specified Outcome: Foot and Ankle Ability Measure (FAAM)
Description: as for outcome 1
Time Frame: 6-Week Cross-over
Measure: Mean (Standard Deviation); unit: Percentage of function
Arm/Group | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention
Number analyzed (Participants) | 26
Percentage of function
  Activities of Daily Living (21- item) | 56.27 (17.32)
  Sports (7-item) | 16.69 (8.88)

14. Other Pre Specified Outcome: Pain Diary Defense and Veterans Pain Rating Scale (DVPRS)
Description: as for outcome 5
Time Frame: 3-Week Cross-over
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention
Number analyzed (Participants) | 26
units on a scale | 3.11 (2.25)

15. Other Pre Specified Outcome: Pain Diary Defense and Veterans Pain Rating Scale (DVPRS)
Description: as for outcome 5
Time Frame: 6-Week Cross-Over
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention
Number analyzed (Participants) | 26
units on a scale | 3.50 (2.34)

16. Other Pre Specified Outcome: Foot and Ankle Ability Measure (FAAM)
Description: as for outcome 1
Time Frame: 3-month Cross-over
Measure: Mean (Standard Deviation); unit: Percentage of function
Arm/Group | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention
Number analyzed (Participants) | 26
Percentage of function
  Activities of Daily Living (21- item) | 57.00 (17.09)
  Sports (7-item) | 16.11 (7.92)

17. Other Pre Specified Outcome: Pain Diary and Veterans Pain Rating Scale (DVPRS)
Description: as for outcome 5
Time Frame: 3-month Cross-over
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention
Number analyzed (Participants) | 26
units on a scale | 3.65 (2.40)

ADVERSE EVENTS:
Time Frame: All participants were evaluated for adverse events during their participation at each follow-up visits(3 weeks, 6 weeks, 3 months, 3-week cross-over, 6-week cross-over, 3-month cross-over) using a standard questionnaire on the IRB-approved follow-up case report form. From August 11, 2022, to October 31, 2024, 7 serious adverse events and three adverse events were documented during the study period. The events were not related to the research procedure.
Description: All adverse events, regardless of severity were reported to the Principle Investigator. The study overall is considered to be minimal risk for study participants, defined as not substantially above what would be encountered in everyday life including provision of routine medical care for the condition of plantar fasciitis. All adverse events, regardless of severity were reported to the Principal Investigator.
Groups:
- The Usual Care + PBM Group: Participants that were assigned to this group received active treatment with PBM 3 times a week for 3 weeks for a total of 9 treatments.
  Photobiomodulation Therapy (PBMT): Participants received PBMT with the PBM device over the course of three consecutive weeks (three treatments per week). PBM treatments will take approximately 5-10 minutes to administer at each session. Specific treatment parameters were based on measurements of calf, ankle, and foot using pre-calculated treatment tables; participants received 10 J/cm2, 25W output power, and the length of the treatment was dependent on treatment area (size).
  PBMT was administered by a trained member of the study team using the LightForce® XPi therapy laser, provided by LiteCure, LLC/DJO Global (New Castle, DE). The LightForce® XPi therapy laser is an FDA cleared device for the treatment of pain. The trained team members will use the Smart Hand Piece technology, which achieves effective treatments and improves dosing accuracy by assessing the operator's speed and providing real-time visual (red - amber - green light) and sensory feedback.
- The Usual Care + Sham (Placebo) PBM Group: Participants that were assigned to this group received Sham PBM therapy 3 times a week for 3 weeks for a total of 9 treatments. Sham PBM therapy is an inactive harmless treatment that is intended to mimic the active PBM treatment.
  Sham-Photobiomodualtion Therapy (Sham-PBMT): Sham-PBM treatment time was calculated in the same way as the PBM treatment group, with the time of treatment dependent on the size of the treatment area. The sham-PBMT was administered by rolling the massage ball over the plantar surface of the foot and dorsal aspect of the calf in contact with the participants' skin. Because emission of photons at the selected treatment parameters may cause participants in the treatment group to feel warmth, the massage was warmed in the sham-PBMT. The device was turned on, so the red aiming beam will be visible, but the operator did not activate the switch to emit photons.
- The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention: Participants that were decided to cross-over to this group received active treatment with PBM 3 times a week for 3 weeks for a total of 9 treatments.
  Photobiomodulation Therapy (PBMT): Participants received PBMT with the PBM device over the course of three consecutive weeks (three treatments per week). PBM treatments took approximately 5-10 minutes to administer at each session. Specific treatment parameters were based on measurements of calf, ankle, and foot using pre-calculated treatment tables; participants received 10 J/cm2, 25W output power, and the length of the treatment was dependent on treatment area (size).
  PBMT was administered by a trained member of the study team using the LightForce® XPi therapy laser, provided by LiteCure, LLC/DJO Global (New Castle, DE). The LightForce® XPi therapy laser is an FDA cleared device for the treatment of pain. The trained team members used the Smart Hand Piece technology, which achieves effective treatments and improves dosing accuracy by assessing the operator's speed and providing real-time visual (red - amber - green light) and sensory feedback.
Arm/Group | The Usual Care + PBM Group | The Usual Care + Sham (Placebo) PBM Group | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/31 | 3/33 | 2/26
Other Adverse Events (participants affected / at risk) | 1/31 | 2/33 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Usual Care + PBM Group (N=31) | The Usual Care + Sham (Placebo) PBM Group (N=33) | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention (N=26)
Arm Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — At the 6-week follow-up, the participant informed the study team that they injured their arm at work and were hospitalized prior to the follow-up. The participant continues to follow up with the patient care management for the injury.
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — At the 3-week follow-up, the participant reported having an illness and was in quarantine.
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — At 6-week follow-up, participant reported having the flu.
Fluid in the Foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) — The participant had fluid in the foot and continues follow-up with a podiatrist who dis discovered the fluid.
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — At 3-week follow-up, participant reported that they went to ER due to significant amount of back pain. Participant continues to be monitored by the patient care management.
Hand Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — At baseline visit, participant reported having hand surgery. Participant continues recovery follow-up with their provider.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Usual Care + PBM Group (N=31) | The Usual Care + Sham (Placebo) PBM Group (N=33) | The Usual Care + Sham (Placebo) PBM Group With Cross-over to Intervention (N=26)
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — At 3-week follow-up, the participant reported minor increase in foot pain.
Skin reaction to unknown (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — After treatment 1, participant reported abnormal feeling on vein of right hand.
Scar from Dry Needling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — As recorded during baseline, participant continues to have lump at arch location on both feet from dry needling procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT05763381/Prot_SAP_002.pdf
  • Informed Consent Form (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT05763381/ICF_003.pdf